CLINICAL TRIAL: NCT01679197
Title: Clinical Protocol to Investigate the Efficacy of Recombinant Human Leptin (Metreleptin) in Nonalcoholic Steatohepatitis (NASH) or Nonalcoholic Fatty Liver Disease (NAFLD) Associated With Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elif Oral, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCRU 2834; R01DK088114-02 (NIH)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Fatty Liver Disease, Nonalcoholic; Nonalcoholic Steatohepatitis; Lipodystrophy
Keywords: Nonalcoholic fatty liver disease; NAFLD; Nonalcoholic steatohepatitis; NASH; Lipodystrophy; Leptin; Metreleptin; Hypertriglyceridemia; Diabetes mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Lipodystrophy; Hypertriglyceridemia; Diabetes Mellitus | interventions — metreleptin; recombinant methionyl human leptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Metreleptin
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin
  Other Names: (originally A100, recombinant-human-methionyl-leptin

SUMMARY:
This study involves research about an investigational medicine called metreleptin. The reason for this study is to find out how metreleptin can improve non-alcoholic steatohepatitis or nonalcoholic fatty liver disease associated with lipodystrophy, a rare disorder associated with abnormal loss of the body's fat tissue. In this study, metreleptin is considered to be investigational for the treatment of lipodystrophy. Metreleptin will be given via injections under the skin. We plan to continue therapy for a period of one year and evaluate the change in liver disease by a liver biopsy. We will also follow the metabolic parameters (e.g. blood cholesterol, liver function, insulin resistance) and body composition characteristics (e.g. the pattern of fat distribution in the body).

DETAILED DESCRIPTION:
The goal is to test the efficacy of restorative leptin therapy on the degree of hepatic steatosis and on amelioration of pathological features of NASH/NAFLD. In addition, the study will evaluate the impact of leptin therapy on total body insulin sensitivity and lipid levels as well as energy expenditure. In order to accomplish this aim, we now propose an efficacy study with recombinant human leptin therapy in patients with all forms of lipodystrophy who also have NASH/NAFLD.

1. AIM 1: To determine the efficacy of leptin in promoting amelioration of body composition, hepatic steatosis and histopathological scores in patients with all forms of lipodystrophy and NAFLD/NASH. We will conduct a 1 year, open-label study, to assess the metabolic effects of recombinant human leptin (METRELEPTIN, AztraZeneca, Wilmington, DE). The primary outcome measure will be NASH scores. We will also explore body weight, insulin sensitivity, glucose and lipid control, body composition, and free fatty acid levels.
2. AIM 2: To Investigate molecular effects of leptin therapy. In parallel to our preliminary studies, gene expression will be performed on individuals participating in Aim 1 at baseline and following 1 year of leptin. We will combine this with measures of liver metabolite levels to provide novel insights into alterations in metabolism that occur secondary to leptin therapy. We will also measure plasma metabolites at baseline and after 2 (optional), 24 and 48 weeks of therapy to assess the dynamic changes induced by leptin and correlate these changes with phenotypic measures.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female ≥ 5 years old at baseline.
* Is male, female not of childbearing potential, or meets all the following criteria if female of childbearing potential (including perimenopausal women who have had a menstrual period within one year):

  * Not breastfeeding
  * Negative pregnancy test result (human chorionic gonadotropin, beta subunit [βhCG]) at baseline (not applicable to hysterectomized females).
  * Must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate when use consistently and correctly, such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire duration of metreleptin treatment.
* Has physician-confirmed lipodystrophy as defined by evidence of generalized (whole body) or partial (limbs) loss of body fat outside the range of normal variation.
* Alcohol consumption of less than 40 grams/week.
* A liver ultrasound confirming non-alcoholic fatty liver disease, or previous liver biopsy confirming NASH status.
* If ≥ 18 years of age, is able to read, understand and sign the U of M IRBMED approved informed consent form (ICF), communicate with study physician and study team, understand and comply with protocol requirements.
* If < 18 and ≥ 7 years of age, is able to read, understand and sign the appropriate U of M IRBMED approved assent form and has a parent or legal guardian that is able to read, understand and sign the ICF.
* If < 7 and ≥ 5 years of age or unable to read, the appropriate assent form must be explained to the child.
* If previously treated with thiazolidinediones or Vitamin E, stable dose of these medications for at least 3 months.

Exclusion Criteria:

* Presence of advanced liver disease (as evidenced by abnormal synthetic function, abnormal PT or albumin).
* Evidence of other etiologies of viral hepatitis.
* Presence of clinically significant hematologic abnormalities (such as neutropenia and/or lymphadenopathy).
* Presence of HIV infection.
* Very poorly controlled diabetes; HbA1c >10%
* Inability to give informed consent.
* Presence of ESRD, any type of active cancer, or >class 2 congestive heart failure ((New York Heart Association Functional Classification System), based on medical history and physical examination.
* Active infection (may be transient).
* Has known allergies to E. coli-derived proteins or hypersensitivity to any component of metreleptin treatment.
* Any other condition in the opinion of the investigators that may impede successful data collection.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-10-08 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Akinci B, Subauste A, Ajluni N, Esfandiari NH, Meral R, Neidert AH, Eraslan A, Hench R, Rus D, McKenna B, Hussain HK, Chenevert TL, Tayeh MK, Rupani AR, Innis JW, Mantzoros CS, Conjeevaram HS, Burant CL, Oral EA. Metreleptin therapy for nonalcoholic steatohepatitis: Open-label therapy interventions in two different clinical settings. Med. 2021 Jul 9;2(7):814-835. doi: 10.1016/j.medj.2021.04.001. Epub 2021 May 12. PMID 35291351
- [Derived] Meral R, Malandrino N, Walter M, Neidert AH, Muniyappa R, Oral EA, Brown RJ. Endogenous Leptin Concentrations Poorly Predict Metreleptin Response in Patients With Partial Lipodystrophy. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1739-e1751. doi: 10.1210/clinem/dgab760. PMID 34677608

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 23
Completed | 19
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.35 (15.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 22
  African American | 1
  Asian | 0
  Native American | 0
  Unknown | 0
  Decline to answer | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Liver Histopathology
Description: Primary outcome will be the total non-alcoholic steatohepatitis (NASH) score read histopathologically from the liver biopsy samples. This outcome measure quantifies the severity of fatty liver disease. At baseline and at the end of the year, patients have undergone a transcutaneous liver biopsy and the specimens were graded for the severity of non-alcoholic fatty liver disease (NAFLD)/non-alcoholic steatohepatitis (NASH) pathology. Histological features of NAFLD/NASH were scored using the validated NASH-CRN (NASH Clinical Research Network) scoring system. This scoring system is the total of 4 subscales: steatosis (0-3), lobular inflammation (0-3), hepatocellular ballooning (0-2) and fibrosis (0-4), which are evaluated semi-quantitatively. The total scale range for this scoring system is 0-12, with 0 representing no features of fatty liver disease, and 12 representing the highest degree of fatty liver disease.
Time Frame: 1 year
Population: The number of participants analyzed at month 12 differs from the overall number analyzed at baseline because 4 participants dropped from the study before their month 12 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 23
units on a scale
  Baseline | 6 (2)
  Month 12: number analyzed (Participants) | 19
  Month 12 | 5 (2)

2. Secondary Outcome: Liver Fat by MRI and MR Spectroscopy
Description: All enrolled patients will have a baseline MRI of the liver to evaluate liver volume and liver fat. For determination of hepatic fat content by MRI and MR spectroscopy in patients, a series of out-phase and in-phase MRI at multiple flip angles are used. By combination of out-phase and in-phase MRI at multiple flip-angles and TE times, relaxation-time effects can be removed to yield quantitative intra-hepatic (and other organs') fractional fat content throughout the liver in a few breath-hold intervals.
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %fat
Arm/Group | Treatment
Number analyzed (Participants) | 23
%fat
  Baseline | 19.19 (11.11)
  Month 12: number analyzed (Participants) | 19
  Month 12 | 13.47 (9.02)

3. Secondary Outcome: Liver Function Tests
Description: AST and ALT are the liver function tests. We are reporting the liver function tests where the treatment group arm would normally be listed, though, we are looking at the same single arm population of 23 participants who received treatment in this study.
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Liver Function AST | Liver Function ALT
Number analyzed (Participants) | 23 | 23
IU/L
  Baseline | 41.52 (27.46) | 53.22 (37.03)
  Month 12: number analyzed (Participants) | 19 | 19
  Month 12 | 30.37 (14.04) | 36 (22.84)

4. Secondary Outcome: Fasting Lipids
Description: Cholesterol, triglycerides, HDL cholesterol, and LDL together make up the lipid profile and must be reported together. We are reporting the lipid profile where the treatment group arm would normally be listed, though, we are looking at the same single arm population of 23 participants who received treatment in this study.
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Cholesterol, Total mg/dL; Triglycerides mg/dL; HDL Cholesterol mg/dL; LDL mg/dL: Lipid measurement
Arm/Group | Cholesterol, Total mg/dL | Triglycerides mg/dL | HDL Cholesterol mg/dL | LDL mg/dL
Number analyzed (Participants) | 23 | 23 | 23 | 23
mg/dL
  Baseline | 256.91 (136.87) | 1057.48 (1744.89) | 35.83 (11.01) | 95.39 (48.30)
  Month 12: number analyzed (Participants) | 19 | 19 | 19 | 19
  Month 12 | 189.11 (64.73) | 478.47 (790.85) | 33.42 (6.41) | 95.95 (32.64)

5. Secondary Outcome: Fasting Glucose
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 23
mg/dL
  Baseline | 178.91 (82.36)
  Month 12: number analyzed (Participants) | 19
  Month 12 | 163.53 (66.79)

6. Secondary Outcome: Body Weight
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment
Number analyzed (Participants) | 23
kg
  Baseline | 77.2 (21.4)
  Month 12 | 75.0 (23.1)

ADVERSE EVENTS:
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 7/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=23)
Left shoulder pain, atypical chest pain (Cardiac disorders) | 1 (1)
Granulomatous tissue reaction (Immune system disorders) | 1 (1)
Bronchial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall, hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Transient ischemic attack vs. cerebrovascular attack vs. complicated migraine (Nervous system disorders) | 1 (1)
Epigastric pain, mild chest pain (Gastrointestinal disorders) | 1 (1)
Secondary diabetes mellitus with keatoacidosis (Metabolism and nutrition disorders) | 1 (1)
Bell's palsy left side weakness (Nervous system disorders) | 1 (1)
UTI abdominal pain (Renal and urinary disorders) | 1 (1)
Rectal prolapse surgery (Surgical and medical procedures) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=23)
Hypoglycemia (Blood and lymphatic system disorders) | 7 (12)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (General disorders) | 2 (2)
Upper respiratory tract infection (Immune system disorders) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Urinary tract infection (Renal and urinary disorders) | 2 (3)
Fall (Musculoskeletal and connective tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (General disorders) | 3 (4)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abdominal pain/discomfort (Gastrointestinal disorders) | 3 (3)
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Cold/Flu-like symptoms (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No